CLINICAL TRIAL: NCT05942313
Title: Predicting and Preventing Adverse Maternal and Child Outcomes of Opioid Use Disorder in Pregnancy
Status: Recruiting | Type: Observational
Sponsor: Ilana Hull (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); OpalGenix, Inc (Industry)
Responsible Party: Sponsor-Investigator, Ilana Hull, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: STUDY23010043; 1R43DA058430-01 (NIH)
Record Dates: First submitted 2023-07-03; First posted 2023-07-12 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Opioid Use Disorder; Pregnancy Related
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Genotyping will be examining CYP2B6, CYP2D6, CYP3A4, OPRM1, OPRK1, ABCB1, FAAH, OCT1, COMT, ABCC3, ADRB2, PNOC and other genes using a comprehensive (1500 genes) Thermo Fisher PharmacoScan panel and OPRM1 epigenetic analyses using Infinium MethylationEPIC kit at College of American Pathologists (CAP) and Clinical Laboratory Improvement Amendments (CLIA) accredited UPMC Genome Center (UGC) and preprocessed as we previously published. Other significant genes and epigenetic associations will be pursued in future genome-wide analysis studies. Infant blood samples will be no more than 3ml/kg in total volume.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pregnant women with Opioid Use Disorder (OUD): This study will enroll 100 pregnant women with OUD at UPMC with its high volumes
  Interventions: Drug: Buprenorphine/ Methadone exposure

INTERVENTIONS:
Drug: Buprenorphine/ Methadone exposure — Validate candidate genes- and prenatal opioid exposure- related maternal relapse and NOWS outcome associations in pregnant women and their newborns.
  Other Names: Opioid Use Disorder

SUMMARY:
This study will be a 12-month prospective, genotype-blinded longitudinal observational study with current standard of clinical care. This study will enroll 100 pregnant women with OUD at UPMC Hospitals with its high volumes. Because of the observational nature of the study, the anticipated dropout rate will be ≤ 20%. Investigators expect the effective sample size of evaluable patients will be 200 with longitudinal data.

DETAILED DESCRIPTION:
Background: 7% of pregnant women in the U.S. use opioids and 21% of these women report misuse, making opioid use disorder (OUD) a major public health concern during pregnancy. The number of infants born with prenatal opioid exposure, neonatal opioid withdrawal syndrome (NOWS) and costly prolonged hospitalization has increased exponentially. The opioid epidemic is further worsened by the ongoing COVID-19 pandemic. Despite medication treatment for OUD with buprenorphine (BUP) or methadone (METH), these pregnant women continue to be at high risk for early relapse, polysubstance use, and depression. These infants are at risk for not only immediate NOWS and also poor long-term neurodevelopmental and behavioral outcomes. Genetic factors influence 30-60% of opioid adverse events (AEs). In pregnant women on medication management for OUD, and infants receiving opioids for NOWS treatment there is variability in dose required to prevent withdrawal symptoms and craving, likely related to physiological alterations, upregulation of metabolic and biological pathways, determined in part by opioid pharmacogenomics. Investigators have shown that in children and adults, opioid related poor clinical outcomes are related to opioid receptor genetic variations and resulting variations in their metabolism. Maternal depression and anxiety increase the risks for OUD, maternal relapse, NOWS and negatively impact pregnant women and their children. Thus, there is an urgent and unmet clinical need for a reliable tool to proactively predict maternal relapse, NOWS, and improve the safety of pregnant women with OUD and their children.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with OUD and their infant
* Currently on BUP/METH for OUD
* Enrolled in prenatal opioid maintenance program
* Age >18 years
* Singleton pregnancy
* Planned delivery at UPMC's Magee Womans Hospital
* Positive opioid urine screen results

Exclusion Criteria:

* Serious maternal medical illness as deemed by the PI that would make it challenging to comply with study procedures
* HIV or AIDS
* Known major fetal congenital abnormalities

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be a 12-month prospective, genotype-blinded longitudinal observational study with current standard of clinical care. This study will enroll 100 pregnant women with OUD at UPMC with its high volumes. Because of the observational nature of the study, the anticipated dropout rate will be ≤ 20%. We expect the effective sample size of evaluable patients will be 200 with longitudinal data.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of maternal opioid relapse | Measured from enrollment to 3-months post delivery
  Measured via binary response, yes/no
Incidence of NOWS | Measured at delivery
  Clinical definition of NOWS: Substance withdrawal encompasses a continuum of variable clinical expression from neonate to neonate; the diagnosis is not limited only to neonates who require pharmacotherapy. Incidence of NOWS measured by binary response, yes/no

SECONDARY OUTCOMES:
Severity of Maternal Opioid Relapse | Measured from enrollment to 3-months post delivery
  Severity of maternal opioid relapse measured by requirement of medical treatment (binary response, yes/no)
Severity of NOWs | Measured at delivery
  Severity of NOWs measured by the need for >3 days of hospital stay (binary response, yes/no)

CONTACTS AND LOCATIONS:
Overall Officials: Ilana Hull, MD, Principal Investigator — Univrsity of Pittsburgh / UPMC Magee Womens Hospital
Locations (1):
- UPMC Magee-Womens Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
We intend to share data that is generated from the grant at the earliest opportunities throughout this research project in counsel with our intellectual property lawyers. The details of the risk prediction algorithms will remain proprietary and will be protected as a trade secret.
Supporting Information: CSR
Time Frame: Data will become available after completion of the two-year enrollment period.
Access Criteria: This information will be held in a commercial cloud-based data portal with a password and encrypted security, such as commercial sources BOX, Dropbox, Engnyte, and Sharepoint. Access to the electronic portal will only be provided after the receiving party has signed a confidentiality agreement. The data will not be downloadable but rather only allow for viewing from the cloud-supported site. This is the process used during corporate due diligence in determining the potential to invest and is an industry-accepted approach. This approach will be used for potential investors and additional collaborators on future projects.